CLINICAL TRIAL: NCT03161106
Title: To Assess Efficacy of Nutritional Therapy in Secondary Prophylaxis of Hepatic Encephalopathy Versus Lactulose in Patients With Liver Cirrhosis- A Randomised Controlled Trial
Brief Title: To Assess Efficacy of Nutritional Therapy in Secondary Prophylaxis of Hepatic Encephalopathy Versus Lactulose in Patients With Liver Cirrhosis.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-12
Record Dates: First submitted 2017-05-08; First posted 2017-05-19 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-06

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Nutritional Status; Lactulose; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrional Therapy Group (Experimental): Nutritional group- Protein of 1.5 gm/kg thrice daily for 6 months
  Interventions: Dietary Supplement: Nutrition
- Lactulose Group (Active Comparator): Lactulose - 20 mL thrice daily (maximum) for 6 months
  Interventions: Drug: Lactulose; Dietary Supplement: Diet

INTERVENTIONS:
Dietary Supplement: Nutrition — Nutrional group-30 kcal/kg with 1.5 grm protein with protein supplements
  Arms: Nutrional Therapy Group
Drug: Lactulose — Lactulose plus diet consumed by patient
  Arms: Lactulose Group
Dietary Supplement: Diet — Protein Powder 15 to 20 gm/meal/day
  Arms: Lactulose Group

SUMMARY:
The study will be conducted on patients attending /admitted to Department of Hepatology from April 2017 to December 2018 at ILBS, New Delhi .

Clinical, anthropometric and biochemical assessment will be done by candidate, co-supervisors and supervisor. Patients in treatment group will receive nutritional therapy in the form of 30-kcal/kg/day and 1.5gm/kg/day protein with supplements. Other patients will continue diet that they were receiving before along with lactulose. Previous treatment and prophylaxis of variceal bleed any (endoscopic variceal ligation or beta blocker) will be continued as before. All subjects will be followed up every month for treatment compliance and for development of any complications.

ELIGIBILITY:
Inclusion Criteria:

1. Liver cirrhosis (Child B or Child C class)
2. Age between 18-60 years
3. History of recovery from episodeof overt hepatic encephalopathy (West-Haven grade 1 and above) in last 12 months.

Exclusion Criteria:

1. Evidence of overt hepatic encephalopathy at the time of enrollment
2. History of taking lactulose, rifaximin, neomycin, metronidazole, L-Ornithine L-Aspartate or probiotics in past 7 days
3. Alcohol intake during past 6 weeks
4. Receiving secondary prophylaxis for spontaneous bacterial peritonitis
5. Previous transjugular intrahepatic portosystemic shunts or shunt surgery
6. Significant comorbid illness such as heart, respiratory or kidney failure, and neurological disease such as Alzheimer's disease, Parkinson's disease and non hepatic metabolic encephalopathies
7. Receiving psychoactive drugs, promotility and hypomotility drugs
8. Hepatocellular carcinoma
9. Electrolyte abnormality (Serum sodium <125meq/L or serum potassium <2.5meq/L)
10. Intercurrent infection such as spontaneous bacterial peritonitis
11. Patients of acute on chronic liver failure (ACLF).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients develop hepatic encephalopathy in both groups | 6 Months

SECONDARY OUTCOMES:
Improvement in health related quality of life over 6 months | 6 Months
  Improvement will be defined on the basis of HRQOL (Health Related Quality of Life Index).
Improvement in anthropometry parameters (mid arm circumference, triceps skin fold thickness, hand grip), skeletal muscle mass, body fat mass, percent body fat,BMI over 6 months | 6 Months
  Improvement will be measured by dexa scan , C T scan and by measuring mid arm circumference, triceps skin fold thickness, hand grip
Time taken for first breakthrough episode of overt hepatic encephalopathy | 6 Months
Time to first overt hepatic encephalopathy-related hospital admission | 6 Months
Mortality over 6 months | 6 Months
Changes in serum cytokines (IL-1,6,10,18,TNF,Endotoxins,myostatin levels) | 6 Months
Changes in Stool microbiota for 20 patients | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No